CLINICAL TRIAL: NCT01548872
Title: Comparison of the Effects of Crystalloid Cardioplegia and HTK Solution for Postoperative Troponin-I and CK-MB Levels After Pediatric Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Selim Kuslu, Anesthesiology Resident, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KA/11-152
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Myocardial Injury
Keywords: HTk solution; Cardioplegia; myocardial protection; pediatric cardiac surgery
MeSH Terms: interventions — Bretschneider cardioplegic solution; potassium cardioplegic solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- crystalloid cardioplegia solution (Active Comparator): After aortic cross clamp 30ml/kg will be administered
  Interventions: Drug: crystalloid cardioplegia solution
- HTK solution (Active Comparator): After aortic cross clamp 50ml/kg will be administered
  Interventions: Drug: HTK solution

INTERVENTIONS:
Drug: HTK solution — 50 ml/kg bolus in 2 minutes
  Arms: HTK solution
Drug: crystalloid cardioplegia solution — 30 ml/kg bolus in two minutes
  Arms: crystalloid cardioplegia solution

SUMMARY:
The purpose of this study is to compare two different cardioplegia solutions effect on postoperative Troponin-I and CK-MB levels after pediatric cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective pediatric cardiac surgery
* Patients written informed consent for study participation

Exclusion Criteria:

* redo surgery
* allergy to study drugs
* unstable blood pressure before cardiac surgery

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
myocardial protective effect of HTK solution | postoperative 48 hours
  to detect %33 difference in Troponin-I levels 4 hours postoperatively

SECONDARY OUTCOMES:
hemodynamic and respiratory data | postoperative 48 hours
  arterial pressures, heart rate,blood gas analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Faculty of Medicine, Ankara, Çankaya, Turkey (Türkiye)